CLINICAL TRIAL: NCT03653741
Title: Effects of Perampanel on Neurophysiology Test Perimeters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1704018150
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Intervention Model Description: 12 healthy males will undergo testing, then receive the drug intervention, followed by blood draw and testing again
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Healthy males (Experimental): healthy males will undergo EEG, VEP, BAER, and SEP testing, then take a single dose of Perampanel 6 MG pill (intervention), then have blood drawn and undergo the 4 tests mentioned previously for a second time
  Interventions: Drug: Perampanel 6 MG

INTERVENTIONS:
Drug: Perampanel 6 MG — Perampanel is a drug approved and marketed in the USA for the treatment of epilepsy to prevent recurrent seizures. In a previous study, healthy volunteers have tolerated a single dose of perampanel at 6 mg quite well.
  Other Names: perampanel

SUMMARY:
This is a study to evaluate the effects of perampanel, a FDA approved drug for epilepsy, on commonly performed neurophysiology tests: electroencephalogram (EEG), somatosensory evoked potential (SEP), brainstem auditory evoked potential (BAEP), and visual evoked potential (VEP). Many other drugs used in the treatment of epilepsy have been shown to affect the results of these test but no one has yet examined if perampanel affects these tests. The investigators plan to recruit 12 healthy normal male subjects. All subjects will have VEP, SSEP, EEG, and BAER performed before and 1 hour (when Cmax is reached) after receiving 6mg of oral perampanel. Subjects will also receive a blood draw 1 hour after ingestion of perampanel for serum perampanel level. In a previous study done at another institution, healthy volunteers have tolerated a single dose of perampanel at 6 mg quite well. There is no placebo nor randomization. Subject's participation concludes after completion of post-perampanel ingestion neurophysiology tests.

DETAILED DESCRIPTION:
The study drug used in this research study is perampanel, an FDA approved medication for the treatment of seizures. The study is being done to examine whether the study drug affects the following non-invasive tests of brain activity: electroencephalogram (EEG), visual evoked potential (VEP), brainstem auditory evoked potential (BAER), and somatosensory evoked potential (SEP). Many anti-seizure drugs have been shown to affect these 4 tests. Anti-seizure medications such as phenytoin, carbamazepine, and oxcarbazepine have been shown to cause slowing of brain activity on EEGs. To date, there have been no published data on whether perampanel, affects EEG, VEP, SEP, or BAER. The data from this study may help with interpretation of these tests in epileptic patients on perampanel.

The investigators are looking for male participants with no prior chronic medical conditions to partake in this study.

All participants will undergo the following tests as part of the study:

1. EEG: this test monitors the electrical activity of the brain through small, metal disks (electrodes) that are placed on the scalp. The test is painless and after the electrodes are placed, participants will be asked to lay down as brain activity is monitored.
2. VEP: this test is similar to the EEG in that electrodes will be placed on the back of the head to monitor brain electrical activity. This test looks specifically at what is happening in the part of the brain that responds to vision, so during the test participants will be shown visual stimuli like a bright light or image on a screen to stimulate brain activity.
3. BAER: this test is similar to the EEG in that electrodes will be placed on participant's head to monitor brain electrical activity. This test looks specifically at what is happening in the part of the brain that responds to sound, so during the test, different sounds will be played to stimulate brain activity.
4. SEP: this test is similar to the EEG in that electrodes will be placed on participant's head to monitor brain electrical activity. This test looks specifically at what is happening in the part of the brain that responds to touch and body sensations, so electrodes will also be placed on the arms and legs to stimulate that area with an electric pulse. This electrical stimulation can cause mild discomfort but is generally well tolerated. Participants may feel muscles twitch when the electrical stimulation is given.

These tests are non-invasive and done routinely in the evaluation of neurologic diseases. They are well tolerated and have no long term side effects.

Following the completion of the four tests, participants will take a single dose of 6mg pill of perampanel:

Perampanel is a drug approved and marketed in the USA for the treatment of epilepsy to prevent recurrent seizures. In a previous study, healthy volunteers have tolerated a single dose of perampanel at 6 mg quite well.

Following taking the pill of perampanel, participants will have their blood drawn:

Participants will have their blood drawn approximately 1 hour after ingestion of single dose of perampanel to measure the concentration of the drug in their blood stream. The total amount of blood taken during the study is approximately 40-60 teaspoons.

After the blood draw, participants will repeat the four tests (EEG, VEP, BAER, SEP) as described above.

There is no follow up visit. However, the study physician will be available should participants experience unexpected side effects due to the study. The investigators, physicians, or sponsors may stop the study or take participants out of the study at any time should they judge that it is in participants' best interest to do so. For instance, they may take participants out of the study if they experience a study-related injury or if they are unable to undergo testing. They may remove participants from the study for various other administrative and medical reasons. They can do this without consent.

For trials of drugs, there may be risks. The research doctor will discuss the full extent of diagnostic, procedural, and drug risks with participants. There may be risks which are currently unforeseeable. As with all medications, side effects may occur and there may be additional side effects, including long term effects, which are at present unknown. Therefore, it is important that participants report any adverse reactions to the study doctor immediately.

In the period immediately following the study, participants should use caution when driving or using heavy machinery, since the study drug may cause imbalance, dizziness or fatigue.

Participants should not take perampanel if theyare allergic to any of the ingredients in the tablet.

Serious Side Effects:

Perampanel may cause new or worse aggressive behavior, homicidal thoughts or threats, hostility, anger, anxiety, irritability, being suspicious or distrustful (believing things that are not true), and other unusual or extreme changes in behavior or mood. Extreme behavioral changes have not been seen in a study of only a single dose of perampanel, and it is not expected that participants will develop such behavioral changes. Participants should contact the study doctor immediately should they experience any of the above.

Antiepileptic drugs, including perampanel, may cause suicidal thoughts or actions in a very small number of people, about 1 in 500. Subjects should call their healthcare providers right away if they have any of the following symptoms, especially if they are new, worse, or worrisome: thoughts about suicide or dying, thoughts of self-harm, attempt to commit suicide, new or worse depression, new or worse anxiety, feeling agitated or restless, panic attacks, trouble sleeping (insomnia), new or worse irritability, acting aggressive, being angry or violent, acting on dangerous impulses, an extreme increase in activity and talking (mania), and other unusual changes in behavior or mood. Participants should call the study doctor immediately if they notice any changes in mood, ideas or behavior.

Most common side effects:

Dizziness, fatigue, sleepiness, irritability, falls, nausea, imbalance, gait problems, vertigo, and weight gain.

Less commonly seen side effects:

Headache, anxiety, upset stomach, vomiting, constipation, urinary tract infection, problems with coordination, rash, bruises, muscle pain, blurry vision, swelling of arms/legs, numbness, memory problems, confusion, euphoria, low blood sodium level, increase triglyceride level, skin laceration, pain in extremities, back pain, and head trauma. Though rare, skin laceration, head trauma, pain in extremities, and back pain are possible with this medication due to imbalance and dizziness leading to falls.

Additional Risks:

The U.S Drug Enforcement Agency (DEA) may classify some, but not all, medicines as controlled substances. Perampanel has been classified as schedule III. Medicines in this category have an approved medical use but have potential for abuse, physical dependence, or psychological dependence. The risk is lower compared to drugs in Schedule I and II. Some other anti-epileptic medicines have also been listed as controlled substances.

It is possible that perampanel may interact with other medicines and herbal supplements that participants are taking. Before starting the study, the study doctor will determine that they are not taking anything that can interact with perampanel.

During the collection of blood samples, participants may experience slight discomfort and a small amount of bleeding, discoloration or bruising at the site where the needle was inserted. Clot formation and infections may occur at the puncture site, but this is extremely rare. Fainting may occur during or shortly after having blood drawn. If faintness is experienced, participants should lie down immediately to avoid possible injury caused by falling, and notify the site study staff.

Perampanel does not affect the ability of men to father children.

Risks of the Tests:

For all fours tests (EEG, VEP, BAER, SEP), participants may experience discomfort from the placement of the electrodes on the scalp. Participants may also experience visual discomfort when they are shown bright lights during the VEP, as well as hearing discomfort when they hear sounds during the BAER. Finally, participants may experience brief discomfort during the SEP when electrical stimulus is created by the electrodes on the arms or legs. These electrical shocks are done as part of routine exams in patients with possible nerve damages and are generally well tolerated. There are no long lasting effects from these mild shocks.

Efforts will be made to protect participants' medical records and other personal information to the extent allowed by law. However, the investigator cannot guarantee absolute confidentiality. Records of study participants are stored and kept according to legal requirements and may be part of participants' medical record. Participants will not be identified personally in any reports or publications resulting from this study. Organizations that may request to inspect and/or copy participants' research and medical records for quality assurance and data analysis include groups such as:

* Weill Cornell Medical College and NewYork-Presbyterian Hospital
* The Institutional Review Board (IRB)
* The Office of Human Research Protection (OHRP)
* The Food and Drug Administration (FDA) and/or their representatives
* Eisai, Inc. The results of this study may be presented at meetings or in publications; however, participants' identities will not be disclosed in these presentations.

Biological samples may be collected, processed, and reported as necessary for purposes of the study. In the event anyone involved with this study is exposed to participants' blood or bodily fluids, it blood may be tested for evidence of hepatitis, AIDS, or other infections without participants' further consent. Participants will be notified of the results.

By signing the consent form, participants authorize the study doctor to release participants' study-related records to Eisai, Inc., the FDA, the IRB, or any other regulatory authority. By signing the consent form, participants authorize access to this confidential information. Participants also authorize the release of their medical records to Weill Cornell Medical College and NewYork-Presbyterian Hospital by any other hospitals or institutions where participants might receive medical care of any kind while they are participating in this study.

The investigator will not be charging participants any fees to participate in this study.

Participants or their insurance companies will be charged for continuing medical care and/or hospitalization that is not a part of the research study.

Participants will be compensated 200 dollars in cash within 2 weeks after completing the study.

Participants should not expect anyone to pay them for pain, worry, lost income, or non-medical care costs that occur from taking part in this research study. Participants should expect no compensation or reimbursement for these costs or any risks and anxieties associated with any such follow up care. Participants or their insurance companies will also be charged for any continuing medical care and/or hospitalization that are not a part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18 to 50 years old with a body mass index of 19-29 kg/m2 will be recruited.

Exclusion Criteria:

* Subjects would be excluded if they use recreational drugs and have any neurologic disease, psychiatric condition or any other condition that may affect outcome and risk subject safety. Furthermore, anyone that would not be able to participate in neurophysiology tests will also be excluded. Subject will also be excluded should they take any over the counter medication or consume caffeine or alcohol 12 hours prior to the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chuang, M.D., Principal Investigator — NYP/WCMC
Locations (1):
- Neurophysiology Laboratory, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Males
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Males
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Visual Evoked Potential (P100) Amplitude
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Population: Data wasn't collected
Arm/Group | Healthy Males
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Baseline Visual Evoked Potential (P100) Latency
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Measure: Mean (Full Range); unit: ms
Arm/Group | Healthy Males
Number analyzed (Participants) | 12
ms | 1.81 [-2.325 to 3.125]

3. Primary Outcome: Change in Baseline Brainstem Auditory Evoked Potential (Waves I, III, V) Amplitude
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Population: data was not collected
Arm/Group | Healthy Males
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Baseline Brainstem Auditory Evoked Potential (Waves I, III, V) Latency
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Measure: Mean (Full Range); unit: ms
Arm/Group | Healthy Males
Number analyzed (Participants) | 12
ms | 0.02 [-0.175 to 0.25]

5. Primary Outcome: Change in Baseline Somatosensory Evoked Potential (N20) Amplitude
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Population: data was not collected
Arm/Group | Healthy Males
Number analyzed (Participants) | 0

6. Primary Outcome: Change in Baseline Somatosensory Evoked Potential (N20) Latency
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Measure: Mean (Full Range); unit: ms
Arm/Group | Healthy Males
Number analyzed (Participants) | 12
ms | -0.256 [-0.325 to 0.175]

7. Primary Outcome: Change in Baseline Electroencephalography Background Frequency Content
Time Frame: pre-dose and post-dose of drug intake, 7 hours
Measure: Mean (Full Range); unit: Hz
Arm/Group | Healthy Males
Number analyzed (Participants) | 12
Hz | -0.25 [-2 to 1]

ADVERSE EVENTS:
Time Frame: 7h
Description: Subjects were asked to report any adverse events during the study visit.
Arm/Group | Healthy Males
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Males (N=12)
drowsiness (General disorders) | 3
headache (Nervous system disorders) | 3
vertigo (Nervous system disorders) | 4
fatigue (General disorders) | 1
nausea (General disorders) | 2
dizziness (General disorders) | 3
nystagmus (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT03653741/Prot_002.pdf